CLINICAL TRIAL: NCT00160147
Title: A Randomized, Double-Blind, Placebo-controlled, Efficacy, Safety, and Tolerability Study of Bifeprunox in the Treatment of Elderly Subjects With Psychosis and Behavioral Disturbances Associated With Dementia of the Alzheimer's Type
Brief Title: Treatment of Elderly Subjects With Psychosis and Behavioral Disturbances Associated With Dementia of the Alzheimer's Type
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was discontinued prematurely on 25 February 2008 due to slow enrollment
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S154.3.016; 2005-003475-20
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2009-06

CONDITIONS: Psychosis and Behavioral Disturbances Associated With Dementia of the Alzheimer's Type
MeSH Terms: conditions — Psychotic Disorders | interventions — bifeprunox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bifeprunox
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: bifeprunox — One week titration with dose adjustments
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
This is a 10-week study with bifeprunox and placebo in elderly subjects with psychosis and behavioral disturbances associated with dementia of the alzheimer's type.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dementia of the Alzheimer's type

Exclusion Criteria:

* History of seizure disorder
* Clinically significant electrocardiogram (ECG)
* Clinical or radiological evidence of stroke, vascular dementia or dementia due to substance abuse, or head trauma

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) Total Score | 10 weeks

SECONDARY OUTCOMES:
Adverse events | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (51):
- United States (35):
  - Site 912, Phoenix, Arizona
  - Site 902, Carson, California
  - Site 903, Long Beach, California
  - Site 911, Pasadena, California
  - Site 922, San Marino, California
  - Site 910, Santa Ana, California
  - Site 929, Hamden, Connecticut
  - Site 914, New Britain, Connecticut
  - Site 931, Norwalk, Connecticut
  - Site 901, Miami, Florida
  - Site 907, North Miami, Florida
  - Site 933, Orange City, Florida
  - Site 934, Atlanta, Georgia
  - Site 917, Blue Ridge, Georgia
  - Site 925, Newnan, Georgia
  - Site 904, New Orleans, Louisiana
  - Site 905, Shreveport, Louisiana
  - Site 906, Shreveport, Louisiana
  - Site 919, Bedford, Massachusetts
  - Site 923, Boston, Massachusetts
  - Site 942, Flowood, Mississippi
  - Site 927, St Louis, Missouri
  - Site 930, St Louis, Missouri
  - Site 940, St Louis, Missouri
  - Site 941, Olean, New York
  - Site 921, Staten Island, New York
  - Site 909, Cincinnati, Ohio
  - Site 908, Oklahoma City, Oklahoma
  - Site 916, Oklahoma City, Oklahoma
  - Site 935, Philadelphia, Pennsylvania
  - Site 932, Humboldt, Tennessee
  - Site 936, Austin, Texas
  - Site 928, Dallas, Texas
  - Site 913, Williamsburg, Virginia
  - Site 918, Waukesha, Wisconsin
- Czechia (5):
  - Site 803, Litoměřice
  - Site 802, Lnáře
  - Site 804, Prague
  - Site 805, Škvorec
  - Site 801, Tábor
- Estonia (2):
  - Site 807, Viljandimaa
  - Site 806, Voru Maakond
- Israel (6):
  - Site 812, Bat Yam
  - Site 808, Beer Yaakov
  - Site 811, Hadera
  - Site 816, Pardes Hana
  - Site 810, Rehovot
  - Site 809, Tirat HaCarmel
- Poland (3):
  - Site 814, Choroszcz
  - Site 813, Gdansk
  - Site 815, Torun